CLINICAL TRIAL: NCT01171378
Title: Single Arm NCRI Feasibility Study of CHOP in Combination With Ofatumumab in Induction and Maintenance for Patients With Newly Diagnosed Richter's Syndrome
Brief Title: Study of Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone (CHOP) With Ofatumumab in Patients With Richter's Syndrome
Acronym: CHOP-OR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: GlaxoSmithKline (Industry); Cancer Research UK (Other); Oxford University Hospitals NHS Trust (Other); NCRI CLL Subgroup (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_018; OFT113560 (Other Grant/Funding Number: Funder: GlaxoSmithKline); 2009-016459-23 (EudraCT Number)
Record Dates: First submitted 2010-07-22; First posted 2010-07-28 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Richter's Syndrome
Keywords: Richter's Syndrome; High-grade transformation in patients with B cell chronic lymphocytic leukemia; Feasibility; Ofatumumab Induction and maintenance; CHOP; CHOP-0; CHOP-OR; Non Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Other): Single arm study
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — 1000mg vials (50ml @ 20mg/ml), or 100mg vials (5ml @20mg/ml), to be given as an Intravenous (IV) infusion.
  Ofatumumab will be infused intravenously on day 1 (300 mg), day 8 (1000 mg) and day 15 (1000mg) in the first cycle, followed by infusions every 3 weeks of 1000 mg on the first day of each cycle for a total of 6 cycles. Maintenance treatment will start 4 weeks after day 1 of cycle 6 in week 20 and consists of six infusions of ofatumumab every 8 weeks
  Other Names: Arzerra

SUMMARY:
The purpose of this study is to evaluate Ofatumumab in combination with CHOP (cyclophosphamide, hydroxydaunorubicin (doxorubicin), Oncovin (vincristine), and prednisone/prednisolone, the standard chemotherapy treatment) in induction and maintenance treatment of Richter's Syndrome. This study aims to evaluate the overall response rate to CHOP-O (CHOP in combination with Ofatumumab) according to the Revised Response Criteria for Malignant Lymphoma. The hypothesis would be that treatment with CHOP-O for Richter's Syndrome (RS), shows a difference in overall survival (more people living longer), when compared with the standard treatment of CHOP-R (CHOP chemotherapy plus Rituximab).

DETAILED DESCRIPTION:
Richter's Syndrome (RS) is a high-grade transformation that occurs in 5-15% of patients with B cell chronic lymphocytic leukaemia (B-CLL). RS is a complication of B-CLL in which the leukemia changes into a fast-growing diffuse large B cell lymphoma (DLBCL). The pathogenesis (mechanism by which the disease is caused) of RS is poorly understood and predictors of transformation and response to treatment are unknown. Management of RS remains unsatisfactory; the mean overall survival of patients treated with conventional chemo-immunotherapy such as CHOP-R is 8 months from the end of treatment.

CHOP is the acronym for a chemotherapy regimen, cyclophosphamide, hydroxydaunorubicin (doxorubicin), Oncovin (vincristine), and prednisone/prednisolone) and the R stands for the monoclonal antibody, Rituximab. Ofatumumab, a next generation monoclonal anti CD20 antibody, has proven single agent activity in relapsed/refractory B-CLL and other non-Hodgkin lymphomas. In addition, it has shown a favourable safety profile in the maintenance setting.

Therefore, we propose to evaluate Ofatumumab in combination with CHOP in induction and maintenance treatment of patients with RS.

The primary objective of the study will be to evaluate overall response rate (ORR) to CHOP-O (CHOP chemotherapy plus Ofatumumab) according to the Revised Response Criteria for Malignant Lymphoma (Cheson).

Secondary objectives will be feasibility of recruitment, progression free survival and overall survival, the clinical benefit and changes in patient reported outcome measures, safety and tolerability.

This is a multi-centre non-randomised Phase II National Cancer Research Institute (NCRI) feasibility study in 35 patients with newly diagnosed Richter's Syndrome in the UK. CHOP-O will be given for six cycles followed by six cycles of Ofatumumab maintenance treatment every eight weeks and a three months follow-up period. The total duration of recruitment will be 24 months starting from the opening of the first site.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to performing any study-specific procedures
* Patients with B-CLL and newly diagnosed not previously treated and biopsy proven DLBCL Richter's transformation
* Computerized tomography (CT) scan performed within 6 weeks prior to starting treatment.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0, 1, 2 or 3
* Age 18 years and over.

Exclusion Criteria:

* CHOP or CHOP-like anthracycline containing treatment for DLBCL within 6 months prior to registration.
* Known central nervous system (CNS) involvement of B-CLL.
* Any malignancy that requires active treatment with the exception of basal cell carcinoma and non-invasive squamous cell carcinoma.
* Chronic or ongoing active infectious disease requiring systemic treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active hepatitis.
* Subjects meeting any of the following criteria must not be enrolled in the study:
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg (the surface antigen of the Hepatitis-B-Virus). In addition, if negative for HBsAg but HBcAb (Hepatitis B core Antibody) positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded. Consent will be sought prior to any test being performed.
* Clinically significant cardiac disease including unstable angina, uncontrolled congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease.
* History of significant cerebrovascular disease in last 6 months.
* Known Human immunodeficiency virus (HIV) positive.
* Known or suspected hypersensitivity to components of investigational product.
* Patients who have received treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to Visit 2 (start of treatment, cycle 1, day 1).
* Current participation in any other interventional clinical study.
* Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
* Breast feeding women or women with a positive pregnancy test at screening.
* Women of childbearing potential not willing to use adequate contraception during study and for 12 months after last dose of Ofatumumab. Adequate contraception is defined as abstinence, hormonal birth control or intrauterine devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-04; Primary Completion 2015-02 (Actual); Study Completion 2016-04-19 (Actual)

PRIMARY OUTCOMES:
Objective response | Week 20
  Objective response as defined by the revised response criteria for malignant lymphoma (Cheson et al, JCO, Vol 25, No 5, 2007).
  Patients will be classified as responders/non-responders as follows: complete remission (CR), nodular partial remission (nPR) and partial remission (PR) are classified as responders; while stable disease (SD) and progressive disease (PD) are classified as non-responders. Non-evaluable patients will be classified as non-responders.

SECONDARY OUTCOMES:
Overall survival | 72 weeks
  Overall survival where length of survival is defined in whole days as the time from entry into the study until death from any cause. For those who are not observed to die during the course of the trial will be censored at their last known follow-up date.
Progression free survival | 72 weeks
  Progression free survival where length of survival is defined in whole days as the time from entry into the study until lymphoma progression or death from any cause. For those who are not observed to progress or die during the course of the trial will be censored at their last known progression-free follow-up date
Duration of response | 72 weeks
  Duration of response defined in whole days as the time between recorded response to disease progression or death from any cause. Patients will be censored at the date of their last follow-up visit at which the response was assessed.
Time to next DLBCL therapy | 72 weeks
  Time to next DLBCL therapy defined in whole days as the time from the end of study treatment and the start of the next DLBCL therapy other than CHOP in combination with ofatumumab. Patients will be censored at the date of their last follow-up visit at which the further treatment was assessed.
Reduction in Tumour Size | 13, 20 and 72 weeks
  Reduction in Tumour Size will be measured by the absolute value of and percentage change in the sum of products of the diameters of the largest abnormal lymph nodes from screening to post-baseline computerised tomography (CT) scans. CT scans will be complemented by positron emission tomography (PET) scanning in patients with bulky (>5cm) lymphadenopathy from B-CLL.
Patient reported outcomes | Baseline, week 13, week 20, every 2 months until week 72 and at week 72.
  Patient reported outcomes these will be assessed using the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionaire) and the EORTC QLQ-CLL16 at baseline and regular follow-up visits throughout the trial.
Safety | Throughout trial and up to 4 weeks post end of treatment
  Safety - Adverse events (AE) and abnormal clinical and laboratory findings will be collected at all follow-up visits and up to 4 weeks post end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Schuh, MD, PhD, MRCP, FRCPath, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (9):
- United Kingdom (9):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrooke's Hospital, Cambridge
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - Kings College Hospital, London
  - Christie Hospital, Manchester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Eyre TA, Clifford R, Roberts C, Boyle L, Francis A, Schuh A, Dutton SJ. Single arm NCRI phase II study of CHOP in combination with Ofatumumab in induction and maintenance for patients with newly diagnosed Richter's syndrome. BMC Cancer. 2015 Feb 13;15:52. doi: 10.1186/s12885-015-1048-9. PMID 25775024
- See also: Click here for more information about this study: Single arm NCRI feasibility study of CHOP in combination with Ofatumumab in induction and maintenance for patients with newly diagnosed Richter's Syndrome — http://www.octo-oxford.org.uk